CLINICAL TRIAL: NCT07316140
Title: A Prospective Study of Validation of the fullPIERS Model in the Prediction of Adverse Maternal Outcomes in Women With Pre- Eclampsia in Sohag University Hospital
Brief Title: fullPIERS Model in the Prediction of Adverse Maternal Outcomes in Preeclampsia
Acronym: Aprospective
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Abdellah Mohmed, Residant, Sohag University
Other Study IDs: Soh-Med-25-10--12Ms
Record Dates: First submitted 2025-12-13; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Preeclampsia; Fullpairs
Keywords: Fullpairs score; Fullpairs; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients diagnosed with preeclampsia, defined by hypertension (systolic BP diagnosed with preeclampsia, defined by hypertension (systolic BP
  ≥140 mmHg and/or diastolic BP ≥90 mmHg, measured twice more than 4 hours apart after 20 weeks gestation) Proteinuria of at least 0.3 g/dl or ≥300 mg of protein in a 24-hour urine collection Urine albumin-creatinine ratio (ACR) ≥30 mg/mmol, or hypertension with end organ dysfunction after20 weeks gestation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Apredictive formula, fullPIERS (Pre-eclampsia Integrated Estimate of Risk Score), can be used to estimate the risk of suffering an adverse outcome using information obtained within 48 hours of admission with pre-eclampsia. The following information is used, serum creatinine, gestational age, platelet count,

DETAILED DESCRIPTION:
Inclusion criteria Patients diagnosed with preeclampsia, defined by hypertension (systolic BP

≥140 mmHg and/or diastolic BP ≥90 mmHg, measured twice more than 4 hours apart after 20 weeks gestation) Proteinuria of at least 0.3 g/dl or ≥300 mg of protein in a 24-hour urine collection Urine albumin-creatinine ratio (ACR) ≥30 mg/mmol, or hypertension with end organ dysfunction after20 weeks gestation

ELIGIBILITY:
* Inclusion Criteria Female patients diagnosed with preeclampsia. Gestational age ≥ 20 weeks.

Hypertension defined as:

Systolic blood pressure ≥ 140 mmHg and/or Diastolic blood pressure ≥ 90 mmHg, measured on at least two occasions more than 4 hours apart.

Proteinuria defined as:

* 300 mg protein in a 24-hour urine collection or
* 0.3 g/dL on urine analysis. Singleton pregnancy. Exclusion Criteria Patients who do not meet the clinical or laboratory diagnostic criteria of preeclampsia.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female Patients diagnosed with preeclampsia
Study Population: exclude patients who do not meet clinical or laboratory definitions of preeclampsia or related conditions.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Validation of the fullPIERS prediction model for adverse maternal outcomes using logistic regression-derived predicted probabilities | 1year
Evaluate the validity of the fullPIERS model in the prediction of adverse maternal outcomes in women with pre-eclampsia in Sohag Governorate, Egypt. | 1year
  The collected data are then will be used to calculate the predicted probability of adverse outcomes using the fullPIERS logistic regression equation logit(p)=2.68+(-5.41×10-2×gestational age) +1.23×(chest pain or dyspnea)+(-2.71×10 -2×creatinine) .

CONTACTS AND LOCATIONS:
Locations (1):
- Obsetatric and gynacological department at Sohag universtiy hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP
Time Frame: 1year
Access Criteria: http:// uptodate. com